CLINICAL TRIAL: NCT03621280
Title: An Open-label Extension Study of Levoketoconazole (2S,4R-ketoconazole) in the Treatment of Endogenous Cushing's Syndrome
Brief Title: Open-label Treatment in Cushing's Syndrome
Acronym: OPTICS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Cortendo AB (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: COR-2017-OLE
Record Dates: First submitted 2018-05-18; First posted 2018-08-08 (Actual); Results first posted 2025-06-19 (Actual); Last update posted 2025-06-19 (Actual); Status verified 2025-06

CONDITIONS: Cushing Syndrome; Cushing Disease
MeSH Terms: conditions — Cushing Syndrome; Pituitary ACTH Hypersecretion

STUDY DESIGN:
Intervention Model Description: Open-Label Extension Study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Levoketoconazole (Experimental): Levoketoconazole taken twice daily up to 1200 mg daily
  Interventions: Drug: Levoketoconazole

INTERVENTIONS:
Drug: Levoketoconazole — Levoketoconazole up to 1200 mg daily
  Other Names: COR-003

SUMMARY:
This is a long-term, open-label extension study of levoketoconazole in participants with endogenous Cushing's Syndrome.

DETAILED DESCRIPTION:
This is a long-term, open-label extension (OLE) study of levoketoconazole in participants with endogenous Cushing's Syndrome (CS) who have completed one or both parent studies or otherwise potentially qualify for this study, as defined in the eligibility criteria.

ELIGIBILITY:
Key Inclusion Criteria:

1. Completed the Extended Evaluation Phase of Study COR-2012-01 (i.e. M12)
2. Completed the Restoration Phase of Study COR-2017-01 (i.e. RES2)

   NOTE: Participants meeting criteria 1 or 2 above who have had a break in therapy may be eligible only after discussion with the Medical Monitor. If eligible, such participants may require re-establishment of the Therapeutic Dose via titration. All participants who have had a break in therapy should be discussed with the Medical Monitor to determine the starting dose of levoketoconazole. Prior to resuming treatment with levoketoconazole, other therapies for Cushing's Syndrome must undergo an appropriate washout period, with minimum durations as follows:
   * Ketoconazole or metyrapone: 2 weeks;
   * Dopamine agonists: bromocriptine (2 weeks), cabergoline (8 weeks);
   * Octreotide acetate LAR, lanreotide Autogel, pasireotide LAR: 12 weeks;
   * Lanreotide SR: 8 weeks;
   * Octreotide acetate (immediate release) or short-acting pasireotide: 1 week;
   * Mifepristone (RU 486, KORLYM): 4 weeks;
   * Megestrol acetate or medroxyprogesterone acetate (and selected other synthetic progestins): 6 weeks.
3. Currently in a named patient program or other Expanded Access Program receiving levoketoconazole
4. Were levoketoconazole-naïve prior to entry and received early rescue therapy with open-label levoketoconazole in Study COR-2017-01.
5. Achieved a clinically meaningful partial response (with reduction of UFC) in Study COR-2017-01 at dose level 7 or at a maximally tolerated dose of levoketoconazole but did not meet the randomization criteria for Study COR-2017-01 at the end of the Dose Titration and Maintenance Phase when randomization was open.
6. Were levoketoconazole-naïve prior to entry and were enrolled in Study COR-2017-01 in the Dose Titration and Maintenance Phase when randomization was closed. (NOTE: Such subjects must receive at least 1 dose of levoketoconazole before transitioning to this study.)

Key Exclusion Criteria:

* Discontinued levoketoconazole while participating in Study COR-2012-01 or Study COR-2017-01 or a named patient program or other Expanded Access program, due to safety or tolerability concerns or lack of efficacy.
* Scheduled for surgery for treatment of CS or received surgery for treatment of CS within the 6 weeks prior to Screening.
* Treated with mitotane within 6 months prior to enrollment.
* History of malignancy, including adrenal or pituitary carcinomas (other than low-risk, well-differentiated carcinomas of thyroid, breast or prostate that are very unlikely to require further treatment in the opinion of the treating physician, or squamous cell or basal cell carcinoma of the skin).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2019-01-07 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Fredric Cohen, MD, Study Chair — Cortendo AB
Locations (30):
- United States (8):
  - The Center for Diabetes and Endocrine Care, Fort Lauderdale, Florida
  - Emory University, Atlanta, Georgia
  - Washington University School of Medicine, St Louis, Missouri
  - University of New Mexico HSC - HSC Sponsored Projects Office, Albuquerque, New Mexico
  - Columbia University Medical Center, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Cleveland Clinic, Cleveland, Ohio
  - Oregon Health & Science University, Portland, Oregon
- Bulgaria (3):
  - Sveti Georgy University Hospital Clinic of Endocrinology and Metabolic Diseases, Plovdiv
  - Alexandovska University Hospital, Sofia
  - University Specialized Hospital for Active Treatment in Endocrinology, Sofia
- APHM Hôpital de la Conception, Marseille, France
- Greece (2):
  - General Hospital of Athens Evangelismos Department of Endocrinology and Diabete, Athens
  - Hippokration General Hospital Endocrinology and Diabetes Department, Thessaloniki
- Semmelweis Egyetem II. Belgyógyászati Klinika, Budapest, Hungary
- Israel (3):
  - Bnai Zion Medical Center Endocrinology Institute, Haifa
  - Rabin Medical Center, Beilinson Campus, Petah Tikva
  - Tel Aviv-Sourasky Medical Center Institute Endocrinology Metabolism & Hypertension, Tel Aviv
- Italy (5):
  - Clinica Endocrinologia malattie del Metabolismo, Ancona
  - AOU Policlinico G. Martino Sezione di Endocrinologia, Messina
  - Via Sergio Pansini 5 Uni Naples FedericoII Dept of Molecular&Clinical Endocrinology&Oncology, Naples
  - Policlinico Universitario Sant'Andrea, Roma
  - University of Turin, Turin
- Erasmus Medical Center, Rotterdam, Netherlands
- Instytut Centrum Zdrowia Matki Polki, Lodz, Poland
- Romania (3):
  - Institutul National de Endocrinologie C.I. Parhon, Cluj-Napoca
  - Spitalul Clinic Judetean de Urgenta Cluj-Napoca, Cluj-Napoca
  - Spitalul Clinic Judetean Mures, Târgu Mureş
- Spain (2):
  - Hospital Universidad De La Ribera, Alzira
  - Hospital Universitario Ramón y Cajal, Madrid

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Prior to enrolling, participants were required to meet all eligibility criteria including specifications with respect to participation and/or completion of participation in COR-2012-01 and/or COR-2017-01.
Pre-assignment Details: There were 52 potential participants screened for participation in COR-2017-OLE; 51 were eligible for participation and 1 was not eligible for participation, as they failed to achieve a therapeutic dose in COR-2017-01.
Period: Overall Study
Arm/Group | Levoketoconazole
Started | 51
Completed | 24
Not Completed | 27

BASELINE CHARACTERISTICS:
Population: Completers: Participants in COR-2017-OLE were considered having completed the study if they had a Month 36 visit before 01 March 2022 and completed the next scheduled visit (Month 39), if they completed the Month 36 visit after 01 March 2022, or if they completed a scheduled visit within 3 months prior to 31 December 2022.
Groups:
- All Participants: All participants who received at least 1 dose of levoketoconazole in COR-2017-OLE.
Arm/Group | All Participants
Number analyzed (Participants) | 51
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: All Participants: Includes all participants that received at least 1 dose of levoketoconazole in COR-2017-OLE Completers: Includes all participants that received at least 1 dose of levoketoconazole in COR-2017-OLE and met the criteria for study completion prior to 31 December 2022.
  years
    All Participants | 44.1 (11.23)
    Completers: number analyzed (Participants) | 24
    Completers | 48.3 (12.37)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: All Participants: Includes all participants that received at least 1 dose of levoketoconazole in COR-2017-OLE Completers: Includes all participants that received at least 1 dose of levoketoconazole in COR-2017-OLE and met the criteria for study completion prior to 31 December 2022.
  Participants
    All Participants: Female | 40
    All Participants: Male | 11
    Completers: number analyzed (Participants) | 24
    Completers: Female | 19
    Completers: Male | 5
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: All Participants: Includes all participants that received at least 1 dose of levoketoconazole in COR-2017-OLE Completers: Includes all participants that received at least 1 dose of levoketoconazole in COR-2017-OLE and met the criteria for study completion prior to 31 December 2022.
  Participants
    All Participants: American Indian or Alaska Native | 1
    All Participants: Asian | 0
    All Participants: Native Hawaiian or Other Pacific Islander | 0
    All Participants: Black or African American | 3
    All Participants: White | 46
    All Participants: More than one race | 0
    All Participants: Unknown or Not Reported | 1
    Completers: number analyzed (Participants) | 24
    Completers: American Indian or Alaska Native | 0
    Completers: Asian | 0
    Completers: Native Hawaiian or Other Pacific Islander | 0
    Completers: Black or African American | 1
    Completers: White | 23
    Completers: More than one race | 0
    Completers: Unknown or Not Reported | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: All Participants: Includes all participants that received at least 1 dose of levoketoconazole in COR-2017-OLE Completers: Includes all participants that received at least 1 dose of levoketoconazole in COR-2017-OLE and met the criteria for study completion prior to 31 December 2022.
  Participants
    All Participants: Hispanic or Latino | 4
    All Participants: Not Hispanic or Latino | 47
    All Participants: Unknown or Not Reported | 0
    Completers: number analyzed (Participants) | 24
    Completers: Hispanic or Latino | 1
    Completers: Not Hispanic or Latino | 23
    Completers: Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants] — Treated with levoketoconazole: Number of participants from each region that received at least 1 dose of levoketoconazole in COR-2017-OLE.
  Participants
    United States | 10
    Bulgaria | 9
    Israel | 6
    Netherlands | 4
    Greece | 5
    Italy | 6
    Poland | 2
    France | 2
    Romania | 3
    Spain | 2
    Hungary | 2
Weight at COR-2017-OLE Baseline [Mean (Standard Deviation); unit: kg] — Population: All Participants: Includes all participants that received at least 1 dose of levoketoconazole in COR-2017-OLE Completers: Includes all participants that received at least 1 dose of levoketoconazole in COR-2017-OLE and met the criteria for study completion prior to 31 December 2022.
  kg
    All Participants | 80.15 (18.994)
    Completers: number analyzed (Participants) | 24
    Completers | 76.58 (17.127)
BMI at COR-2017-OLE Baseline [Mean (Standard Deviation); unit: kg/m^2] — Population: All Participants: Includes all participants that received at least 1 dose of levoketoconazole in COR-2017-OLE Completers: Includes all participants that received at least 1 dose of levoketoconazole in COR-2017-OLE and met the criteria for study completion prior to 31 December 2022.
  kg/m^2
    All Participants | 29.57 (7.064)
    Completers: number analyzed (Participants) | 24
    Completers | 28.38 (5.962)
Receiving Anti-diabetic Medication at COR-2017-OLE Baseline [Count of Participants; unit: Participants] — Population: All Participants: Includes all participants that received at least 1 dose of levoketoconazole in COR-2017-OLE Completers: Includes all participants that received at least 1 dose of levoketoconazole in COR-2017-OLE and met the criteria for study completion prior to 31 December 2022.
  Participants
    All Participants | 16
    Completers: number analyzed (Participants) | 24
    Completers | 8
Receiving Anti-Hypertensive Medication at COR-2017-OLE Baseline [Count of Participants; unit: Participants] — Population: All Participants: Includes all participants that received at least 1 dose of levoketoconazole in COR-2017-OLE Completers: Includes all participants that received at least 1 dose of levoketoconazole in COR-2017-OLE and met the criteria for study completion prior to 31 December 2022.
  Participants
    All Participants | 33
    Completers: number analyzed (Participants) | 24
    Completers | 17
Receiving Cholesterol-Reducing Medication at COR-2017-OLE Baseline [Count of Participants; unit: Participants] — Population: All Participants: Includes all participants that received at least 1 dose of levoketoconazole in COR-2017-OLE Completers: Includes all participants that received at least 1 dose of levoketoconazole in COR-2017-OLE and met the criteria for study completion prior to 31 December 2022.
  Participants
    All Participants | 8
    Completers: number analyzed (Participants) | 24
    Completers | 6

OUTCOME MEASURES:

1. Primary Outcome: Proportions of Participants With Mean Urinary Free Cortisol (mUFC) Categorization Based on Upper Limit of Normal (ULN)
Description: Proportions of participants with mUFC: 1) Less or equal to the ULN of the reference range, 2) Above the ULN to 1.5x the ULN, and 3) Above 1.5x the ULN.
Time Frame: From parent study Baseline to final study visit or up to a maximum of 3 years, whichever comes first.
Population: The number of participants at each timepoint is based on both the number of participants with evaluable mUFC data at each timepoint and the number of participants remaining in the study at each assessment timepoint.
Measure: Count of Participants; unit: Participants
Arm/Group | All Participants
Number analyzed (Participants) | 51
Participants
  Original Baseline: Less than or equal to ULN | 0
  Original Baseline: Above ULN to 1.5x ULN | 1
  Original Baseline: Above 1.5x ULN | 50
  COR-2017-OLE Baseline: number analyzed (Participants) | 50
  COR-2017-OLE Baseline: Less than or equal to ULN | 26
  COR-2017-OLE Baseline: Above ULN to 1.5x ULN | 12
  COR-2017-OLE Baseline: Above 1.5x ULN | 12
  Month 6: number analyzed (Participants) | 40
  Month 6: Less than or equal to ULN | 20
  Month 6: Above ULN to 1.5x ULN | 10
  Month 6: Above 1.5x ULN | 10
  Month 12: number analyzed (Participants) | 37
  Month 12: Less than or equal to ULN | 15
  Month 12: Above ULN to 1.5x ULN | 11
  Month 12: Above 1.5x ULN | 11
  Month 18: number analyzed (Participants) | 28
  Month 18: Less than or equal to ULN | 16
  Month 18: Above ULN to 1.5x ULN | 6
  Month 18: Above 1.5x ULN | 6
  Month 24: number analyzed (Participants) | 29
  Month 24: Less than or equal to ULN | 18
  Month 24: Above ULN to 1.5x ULN | 5
  Month 24: Above 1.5x ULN | 6
  Month 30: number analyzed (Participants) | 24
  Month 30: Less than or equal to ULN | 15
  Month 30: Above ULN to 1.5x ULN | 3
  Month 30: Above 1.5x ULN | 6
  Month 36: number analyzed (Participants) | 13
  Month 36: Less than or equal to ULN | 7
  Month 36: Above ULN to 1.5x ULN | 3
  Month 36: Above 1.5x ULN | 3

ADVERSE EVENTS:
Time Frame: Up to 3 years; from start of treatment through end of study.
Arm/Group | All Participants
All-Cause Mortality (participants affected / at risk) | 3/51
Serious Adverse Events (participants affected / at risk) | 20/51
Other Adverse Events (participants affected / at risk) | 48/51
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Participants (N=51)
Corona virus infection (Infections and infestations) | 3 (3)
Cellulitis (Infections and infestations) | 1 (1)
Mediastinitis (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1)
Septic shock (Infections and infestations) | 1 (1)
Angina unstable (Cardiac disorders) | 1 (1)
Cardio-respiratory arrest (Cardiac disorders) | 1 (1)
Pericardial effusion (Cardiac disorders) | 1 (2)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pharyngeal haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 3 (3)
Adrenal insufficiency (Endocrine disorders) | 1 (1)
Hyperadrenocorticism (Endocrine disorders) | 1 (1)
Cholecystitis acute (Hepatobiliary disorders) | 1 (1)
Hypertansaminasaemia (Hepatobiliary disorders) | 1 (1)
Aortic dissection (Vascular disorders) | 1 (2)
Essential hypertension (Vascular disorders) | 1 (1)
Ear canal stenosis (Ear and labyrinth disorders) | 1 (1)
Colitis (Gastrointestinal disorders) | 1 (1)
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Presyncope (Nervous system disorders) | 1 (1)
Major depression (Psychiatric disorders) | 1 (1)
Pituitary tumour removal (Surgical and medical procedures) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Participants (N=51)
Corona virus infection (Infections and infestations) | 8 (8) — Does not include the 3 events/participants with corona virus infection that met the criteria for serious.
Upper respiratory tract infection (Infections and infestations) | 5 (8)
Urinary tract infection (Infections and infestations) | 3 (3)
Anaemia (Blood and lymphatic system disorders) | 3 (3)
Palpitations (Cardiac disorders) | 3 (4)
Vertigo (Ear and labyrinth disorders) | 5 (5)
Adrenal insufficiency (Endocrine disorders) | 5 (7)
Nausea (Gastrointestinal disorders) | 17 (26)
Diarrhoea (Gastrointestinal disorders) | 7 (11)
Abdominal pain (Gastrointestinal disorders) | 3 (3)
Abdominal pain upper (Gastrointestinal disorders) | 3 (4)
Dyspepsia (Gastrointestinal disorders) | 3 (3)
Vomiting (Gastrointestinal disorders) | 3 (6)
Fatigue (General disorders) | 10 (13)
Oedema peripheral (General disorders) | 4 (5)
Pyrexia (General disorders) | 4 (4)
Contusion (Injury, poisoning and procedural complications) | 5 (5)
Gamma-glutamyltransferase increased (Investigations) | 4 (5)
Alanine aminotransferase increased (Investigations) | 3 (4)
Hypokalaemia (Metabolism and nutrition disorders) | 12 (15)
Decreased appetite (Metabolism and nutrition disorders) | 3 (4)
Back pain (Musculoskeletal and connective tissue disorders) | 7 (8)
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 (7)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 3 (3)
Myalgia (Musculoskeletal and connective tissue disorders) | 3 (3)
Neck pain (Musculoskeletal and connective tissue disorders) | 3 (3)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 (3)
Headache (Nervous system disorders) | 12 (21)
Dizziness (Nervous system disorders) | 5 (5)
Sciatica (Nervous system disorders) | 3 (4)
Depression (Psychiatric disorders) | 5 (5)
Insomnia (Psychiatric disorders) | 4 (4)
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (5)
Dry skin (Skin and subcutaneous tissue disorders) | 6 (8)
Rash (Skin and subcutaneous tissue disorders) | 5 (6)
Alopecia (Skin and subcutaneous tissue disorders) | 3 (3)
Pruritis (Skin and subcutaneous tissue disorders) | 3 (4)
Hypertension (Vascular disorders) | 14 (20)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The disclosure restrictions aligned with local requirements, allow Sponsor time to submit a multi-center publication after study completion prior to individual site publication. The Sponsor could review results communications before release, request changes and/or removal of confidential information and prohibit communication about trial results for more than 60 days but less than or equal to 6 months from the time submitted for Sponsor review. The Sponsor cannot extend the embargo.

DOCUMENTS (2):
  • Study Protocol (2019-09-23): https://cdn.clinicaltrials.gov/large-docs/80/NCT03621280/Prot_000.pdf
  • Statistical Analysis Plan (2023-02-28): https://cdn.clinicaltrials.gov/large-docs/80/NCT03621280/SAP_001.pdf